CLINICAL TRIAL: NCT01183325
Title: Multicentric Evaluation of the Proceed Ventral Patch for Umbilical and Small Primary Ventral Hernias Less Than 3cm Diameter With One Year Follow-up
Brief Title: Prospective Evaluation of the Proceed Ventral Patch With and Without Laparoscopic Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/291
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Umbilical Hernias; Ventral Hernias
Keywords: Umbilical and small ventral hernias less than 3cm diameter
MeSH Terms: conditions — Hernia, Umbilical; Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proceed Ventral Patch placement (Experimental): Placement of a Proceed Ventral Patch for umbilical and small ventral hernias less than 3cm diameter with and without laparoscopic control
  Interventions: Device: Proceed Ventral Patch placement

INTERVENTIONS:
Device: Proceed Ventral Patch placement — Placement of a Proceed Ventral Patch for umbilical and small ventral hernias less than 3cm diameter with and without laparoscopic control

SUMMARY:
For small (2-3cm) ventral and umbilical hernias the discussion for primary suture repair or the use of mesh continues.

About 5 years ago the Ventralex patch was introduced, which combines a layer of PTFE mesh with a small polypropylene mesh and includes a circular memory ring. Despite the elegance of using this patch, recent experience showed several drawbacks both in design and efficacy (3).

With the recent development of the Proceed Ventral Patch (PVP), new elements have been introduced to overcome some of these issues.

The aim of this study is to evaluate the efficacy of clinical placement of the PVP in the intra-abdominal position in the treatment of small ventral hernias.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Written informed consent
* Umbilical, primary ventral hernias smaller than 3cm diameter

Exclusion Criteria:

* Hernias larger than 3cm
* Recurrence
* Children
* Emergency cases
* Incisional hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of adequately placed patches | At T 0 days

SECONDARY OUTCOMES:
Perioperative morbidity rate | Within 30 days
Pre- and postoperative pain | At T 0 day, T 30 days and T 1 year
Number of patients needed a repositioning of the patch | At T 0 days
Reasons for inadequate positioning | At T 0 days
Number of repositioning necessary | At T 0 days
Complication ratio | At 1 year
Recurrence rate at 1 year | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: Website of University Hospital Ghent — http://www.uzgent.be